CLINICAL TRIAL: NCT07177326
Title: Combination Therapy of Tadalafil 2.5mg Plus Sildenafil 25mg Versus Tadalafil 5 mg Monotherapy for Treatment of Erectile Dysfunction: A Randomized, Placebo-Controlled Double-Blinded Cross-Over Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Khedr, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tadal+Silden VSTadal ED
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Active Comparator): patients recived Tadalafil 2.5 mg + Sildenafil 25 mg.
  Interventions: Drug: Tadalafil 2.5 mg; Drug: Sildenafil 25 mg
- Group2 (Active Comparator): patients recived Tadalafil 5 mg monotherapy
  Interventions: Drug: Tadalafil 5 mg

INTERVENTIONS:
Drug: Tadalafil 2.5 mg — patients recived Tadalafil 2.5 mg daily
  Arms: Group 1
Drug: Sildenafil 25 mg — patients recived Sildenafil 25 mg daily
  Arms: Group 1
Drug: Tadalafil 5 mg — patients recived Tadalafil 5 mg daily
  Arms: Group2

SUMMARY:
Erectile dysfunction (ED) is characterized by the persistent inability to attain or sustain an erection adequate for satisfactory sexual intercourse. As one of the most common male sexual health disorders, ED exhibits a global prevalence of moderate-to-severe cases ranging between 5% and 20% (1). Although erectile dysfunction is not life-threatening, it can substantially impair both physical and psychosocial well-being, exerting a notable negative impact on the quality of life of affected individuals and their partners.

ED is a multifactorial condition associated with vascular, psychological, and, in some cases, idiopathic causes (2). Management strategies encompass lifestyle modification, pharmacotherapy particularly with phosphodiesterase type 5 (PDE5) inhibitors, vacuum erection devices, intracavernosal injections, and surgical options (1). ED frequently coexists with metabolic and cardiovascular disorders and shows a rising incidence with advancing age and the presence of cardiovascular risk factors (2). Both physiological and psychological mechanisms may underlie the condition; psychological etiologies tend to be more prevalent in younger, otherwise healthy individuals (3). The presence of preserved nocturnal erections is a key clinical indicator suggestive of a psychogenic origin of ED (4).

Phosphodiesterase-5 inhibitors (PDE5Is) represent the primary pharmacologic therapy for ED. Currently, seven PDE5Is (avanafil, lodenafil, mirodenafil, sildenafil, tadalafil, udenafil, and vardenafil) are available in varying dosages and formulations. Their efficacy has been consistently demonstrated in randomized controlled trials (5)(6).

Sildenafil exhibits a rapid onset of action, typically beginning 30 minutes after administration, with an effective duration of 4 to 6 hours and a maximum pharmacological activity lasting up to 12 hours (7). While sildenafil is effective in managing erectile dysfunction, discontinuation rates among responders range from 20% to 50% (8). In contrast, tadalafil, a selective and long-acting PDE5 inhibitor introduced in 2003, has a slightly faster onset around 20 minutes and is recommended to be taken at least 30 minutes before sexual activity. Notably, tadalafil has the longest duration of action among PDE5 inhibitors, with effects lasting up to 72 hours. Approximately 52% of patients are able to achieve successful intercourse within 30 minutes of ingestion (9). The purpose of this study is to evaluate the efficacy and safety of Tadalafil 2.5 mg plus sildenafil 25 mg as a combination therapy versus tadalafil 5 mg monotherapy for Treatment of Erectile Dysfunction

ELIGIBILITY:
Inclusion Criteria:

* -Men aged 18-70 years with a clinical diagnosis of erectile dysfunction (ED) for ≥3 months.
* International Index of Erectile Function (IIEF-5) score ≤21.
* Stable sexual relationship for ≥3 months.
* Willingness to adhere to the study protocol and provide informed consent.
* No prior use of PDE5 inhibitors within 4 weeks before enrollment.

Exclusion Criteria:

* -Severe cardiovascular disease (uncontrolled hypertension, recent MI/stroke).
* Hypersensitivity to tadalafil, sildenafil, or any PDE5 inhibitor.
* Severe hepatic/renal impairment (e.g., CrCl <30 mL/min, Child-Pugh C).
* Concomitant use of nitrates, strong CYP3A4 inhibitors (e.g., ritonavir, ketoconazole).
* History of priapism, penile deformities, or radical prostatectomy.
* Major psychiatric disorders affecting compliance.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male only
Enrollment: 142 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Erectile Function (IIEF-5 Score) | 12 week
  Change in Erectile Function (IIEF-5 Score)